CLINICAL TRIAL: NCT01675960
Title: A Phase II, Randomized, Placebo-controlled, Double Blind, Cross-over, Study of the Effects of Gabapentin on Chronic Irritability in Neurologically Impaired Children
Brief Title: Effectiveness of Gabapentin on Chronic Irritability in Neurologically Impaired Children
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: unable to enroll
Sponsor: Gillette Children's Specialty Healthcare (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 112909
Record Dates: First submitted 2012-05-29; First posted 2012-08-30 (Estimated); Results first posted 2019-08-02 (Actual); Last update posted 2019-08-02 (Actual); Status verified 2019-07

CONDITIONS: Neurologically Impaired; Irritable Mood; Signs and Symptoms, Digestive; Sleeplessness; Chronic Pain
Keywords: chronic irritability; chronic pain; Neurologically impaired; gabapentin
MeSH Terms: conditions — Signs and Symptoms, Digestive; Sleep Initiation and Maintenance Disorders; Chronic Pain | interventions — Gabapentin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Gabapentin, then placebo (Experimental): Participants first receive gabapentin 3 times per day, with varying dosing based on the protocol. After 34-38 days, a washout period of 3 days occurs, before then receiving the placebo dose for 32 days.
  Interventions: Drug: Gabapentin; Drug: placebo
- Placebo, then Gabapentin (Experimental): Participants first receive placebo 3 times per day. After 34-38 days, a washout period of 3 days occurs, before then receiving Gabapentin, with varying dosing based on the protocol, for 32 days.
  Interventions: Drug: Gabapentin; Drug: placebo

INTERVENTIONS:
Drug: Gabapentin — The active drug is in a flavored glycerin based solution. The drug will be given orally or through a gastrointestinal tube. Titration up to a stable dose will take 22 days. The total stable dose is 40mg/kg/day. Once 7 days on this dose are finished, children will take 6 days to reduce their dose and begin their 3 day washout period.
  Other Names: Fanatrex; Neurontin; Gabarone; Gralise; Horizant
Drug: placebo — The placebo is a glycerin-based clear solution that is flavored similarly to the commercial product. The placebo will be given orally or through a gastrointestinal tube.

SUMMARY:
This study is a prospective, randomized, double blind, placebo controlled, crossover clinical trial looking at whether gabapentin can provide symptom relief for chronic irritability in neurologically impaired children. The investigators hypothesize gabapentin ins beneficial and safe for children with chronic irritability that persists despite identification and appropriate management of symptom sources.

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled, cross-over study design of the effects of gabapentin on chronic irritability in neurologically impaired children. The study will involve a 22 day medication titration, followed by a 7 day stable dosing period and a 6 day medication taper period. After an additional 3 day washout period, the subject will cross-over to the remaining arm of the study. Subjects will be evaluated for symptoms of chronic pain. Since the subjects are generally non-communicative, the subjects will be evaluated by two questionnaires and the Non-Communicating Children's Pain Checklist-Revised, to be completed by their parent or primary caregiver.

The primary aim is to determine if gabapentin provides symptom relief for chronic irritability in neurologically impaired children.

ELIGIBILITY:
Inclusion Criteria:

* male or female
* 1 month to 16 years of age at enrollment
* neurological impairment defined as subnormal (-2 S.D.) motor and/or cognitive ability from a variety of etiologies
* chronic irritability defined as symptoms suggesting pain to the child's caregiver recurrently over a 4-week of greater time period
* Subject must have an acceptable surrogate capable of giving consent on the subject's behalf

Exclusion Criteria:

* Children with resolved symptoms after treatment of identified sources of pain
* Identified potential source of irritability without adequate trial of appropriate management
* Ketogenic diet
* Renal insufficiency or failure
* Current treatment with gabapentin or pregabalin for another existing condition.

Ages: 1 Month to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2 (Actual)
Dates: Start 2012-04 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Schwantes, MD, Principal Investigator — Gillette Children's Specialty Healthcare
Locations (1):
- Gillette Children's Specialty Healthcare, Saint Paul, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Perquin CW, Hazebroek-Kampschreur AAJM, Hunfeld JAM, Bohnen AM, van Suijlekom-Smit LWA, Passchier J, van der Wouden JC. Pain in children and adolescents: a common experience. Pain. 2000 Jul;87(1):51-58. doi: 10.1016/S0304-3959(00)00269-4. PMID 10863045
- [Background] Breau LM, Camfield CS, McGrath PJ, Finley GA. The incidence of pain in children with severe cognitive impairments. Arch Pediatr Adolesc Med. 2003 Dec;157(12):1219-26. doi: 10.1001/archpedi.157.12.1219. PMID 14662579
- [Background] Houlihan CM, O'Donnell M, Conaway M, Stevenson RD. Bodily pain and health-related quality of life in children with cerebral palsy. Dev Med Child Neurol. 2004 May;46(5):305-10. doi: 10.1017/s0012162204000507. PMID 15132260
- [Background] Stallard P, Williams L, Lenton S, Velleman R. Pain in cognitively impaired, non-communicating children. Arch Dis Child. 2001 Dec;85(6):460-2. doi: 10.1136/adc.85.6.460. PMID 11719327
- [Background] Greco C, Berde C. Pain management for the hospitalized pediatric patient. Pediatr Clin North Am. 2005 Aug;52(4):995-1027, vii-viii. doi: 10.1016/j.pcl.2005.04.005. PMID 16009254
- [Background] Breau LM, Camfield CS, McGrath PJ, Finley GA. Risk factors for pain in children with severe cognitive impairments. Dev Med Child Neurol. 2004 Jun;46(6):364-71. doi: 10.1017/s001216220400060x. PMID 15174527
- [Background] Zangen T, Ciarla C, Zangen S, Di Lorenzo C, Flores AF, Cocjin J, Reddy SN, Rowhani A, Schwankovsky L, Hyman PE. Gastrointestinal motility and sensory abnormalities may contribute to food refusal in medically fragile toddlers. J Pediatr Gastroenterol Nutr. 2003 Sep;37(3):287-93. doi: 10.1097/00005176-200309000-00016. PMID 12960651
- [Background] Hauer JM, Wical BS, Charnas L. Gabapentin successfully manages chronic unexplained irritability in children with severe neurologic impairment. Pediatrics. 2007 Feb;119(2):e519-22. doi: 10.1542/peds.2006-1609. PMID 17272610
- [Background] Breau LM, Camfield C, McGrath PJ, Rosmus C, Finley GA. Measuring pain accurately in children with cognitive impairments: refinement of a caregiver scale. J Pediatr. 2001 May;138(5):721-7. doi: 10.1067/mpd.2001.112247. PMID 11343050
- [Background] Breau LM, McGrath PJ, Camfield CS, Finley GA. Psychometric properties of the non-communicating children's pain checklist-revised. Pain. 2002 Sep;99(1-2):349-57. doi: 10.1016/s0304-3959(02)00179-3. PMID 12237214

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Gabapentin, Then Placebo | Placebo, Then Gabapentin
Started | 2 | 0
Completed | 2 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: There was no one enrolled on Placebo
Groups:
- Total: Total of all reporting groups
Arm/Group | Gabapentin, Then Placebo | Placebo, Then Gabapentin | Total
Number analyzed (Participants) | 2 | 0 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 |  | 2
  Between 18 and 65 years | 0 |  | 0
  >=65 years | 0 |  | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 |  | 0
  Male | 2 |  | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 0 |  | 0
  White | 2 |  | 2
  More than one race | 0 |  | 0
  Unknown or Not Reported | 0 |  | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2 |  | 2

OUTCOME MEASURES:

1. Primary Outcome: Symptom Relief for Chronic Irritability in Neurologically Impaired Children Using Gabapentin.
Description: We will determine whether gabapentin provides symptom relief for chronic irritability in neurologically impaired children, who continue to have irritability even though potential sources may have been identified and treated, or have sources that have not been identified.
Time Frame: Compiled data reviewed at completion or withdrawal from study (3 months from beginning study).
Population: No one was ever enrolled in the placebo arm. The data was never analyzed for this secondary outcome. PI has left the organization therefore analysis will not occur.
Groups:
- Gabapentin: Neurotin
  Gabapentin: The active drug is in a flavored glycerin based solution. The drug will be given orally or through a gastrointestinal tube. Titration up to a stable dose will take 22 days. The total stable dose is 40mg/kg/day. Once 7 days on this dose are finished, children will take 6 days to reduce their dose and begin their 3 day washout period.
- Placebo: Glycerin based clear solution that is flavored similar to the commercial product
  placebo
Arm/Group | Gabapentin | Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Prevalence of Associated Gastrointestinal and Sleep Problems in Neurologically Impaired Children and Improvement Using Gabapentin.
Description: We will attempt to identify gastrointestinal and sleep problems in neurologically impaired children with questionnaires given throughout the study. We hypothesize that gastrointestinal symptoms (feeding intolerance and symptoms associated with gas and bowel movements) and disrupted sleep are frequently associated with chronic irritability and will improve with gabapentin.
Time Frame: Compiled data reviewed at completion or withdrawal from study (3 months from beginning study).
Population: as for outcome 1
Arm/Group | Gabapentin | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected during each contact with the subject after initial drug administration. Patient contacts were scheduled at day 6, 13, 24, 28, 34-37, 38, 44, 51, 62, and 76. SAE still ongoing at end of study period will be followed up on to determine final outcome.
Description: Adverse events are collection on all participants who received at least one dose of intervention, regardless of arm.
Arm/Group | Gabapentin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 1/2 | 0/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gabapentin (N=2) | Placebo (N=2)
Increased sleepiness (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2013-04-26): https://cdn.clinicaltrials.gov/large-docs/60/NCT01675960/Prot_000.pdf
  • Statistical Analysis Plan (2013-04-26): https://cdn.clinicaltrials.gov/large-docs/60/NCT01675960/SAP_001.pdf